CLINICAL TRIAL: NCT04810273
Title: Effect of Progressive Early Mobilization on Functional Recovery in Patients With Moderate-Severe Traumatic Brain Injury: a Single Blind, Randomized Controlled Trial
Brief Title: Effect of Progressive Early Mobilization in Patients With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202012084RIN
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2021-01

CONDITIONS: Early Waking; Trauma; ICU Acquired Weakness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early mobilization (ER) group (Experimental): Participants in the EM group will undergo the progressive early mobilization protocol in the trauma ICU in a manner consistent with the our hospital practice guidelines indicated by the Modified ICU Mobility Scale for progressive mobilization during the ICU stay. EM will be started with in-bed exercises and, if no medical contraindications are present, progressed from sitting in bed with the head tilted >60° to sitting on the edge of the bed to standing (including pre-gait exercises to improve postural stability, static and dynamic balance, and marching on the spot) and, finally, to walking.
  Interventions: Behavioral: Early progressive mobilization
- standard early rehabilitation (SER) group (Active Comparator): Patients in the SER group (Progressive upright positioning protocol) will receive standard physiotherapy including passive range of motion exercises, active exercises, bed mobility, and respiratory therapy during their ICU stays. In the SER group, out-of-bed mobilization (>=Level III in the Modified Trauma ICU Mobility Scale) will be started as soon as possible after ICU discharge but at least Level III (sitting on the edge of bed) above 7 days of onset.
  Interventions: Behavioral: Early progressive mobilization

INTERVENTIONS:
Behavioral: Early progressive mobilization — The goal will be to achieve a mobilization level of at least Level III (sitting on the edge of bed) during the ICU stay (within 7 days).

SUMMARY:
traumatic brain injury (TBI) is a major public health concern worldwide. Patients with moderate-severe TBI have high rates of disability at the acute phase and frequently require protracted rehabilitation with prolonged periods of recovery. Recently, it has been found that the use of progressive early mobilization (EM) protocols for critical trauma patients may minimize the functional declines during intensive care unit (ICU) stays. However, prior early mobilization studies have found that the survivors of moderate-severe TBI often experience a greater incidence of neurological injuries with other organ injury than other critical care patients. No randomized controlled trials thus far have utilized measure the influence or effect of early progressive EM protocols on the functional recovery of moderate-severe TBI patients.

DETAILED DESCRIPTION:
Objective: The goals of this proposed research study are (1) to investigate the feasibility of using a structured progressive EM protocol for patients with moderate-severe TBI in a trauma ICU and (2) The goal is to investigate and compare the intervention effects of a progressive EM protocol (aimed at bringing patients at least to the mobility level-3 of sitting on the edge of bed) in an ICU on short-term and long-term functional abilities in patients with moderate-severe TBI.

ELIGIBILITY:
Inclusion Criteria:

* Expected to stay for at least 72 hours in the ICU,
* >20 years of age with living independently before the onset of critical illness
* relatively stable vital signs with a Glasgow Coma Scale (GCS) score of ≥6
* relatively stable respiratory status (SpO2 >92%, high mechanical ventilator setting: FiO2 ≤60%, and positive end-expiratory pressure ≤10 cmH2O)
* stable cardiovascular system (resting heart rate ≤130 bpm or no use of high-dose vasopressor of more than 0.2 μg kg-1 min-1)

Exclusion Criteria:

* predicted mortality within the next 24 hours
* palliative care
* consistent increase of intracranial pressure (>20 mmHg)
* pregnancy
* uncontrolled seizure
* active bleeding
* ruptured or leaking aortic aneurysm
* development of acute myocardial infarction during ICU stay
* rapid development of degenerative neuromuscular diseases
* contraindication for early walking

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
The total score-change of the Perme ICU Mobility Score | at baseline; at the time of ICU discharge; the time of hospital discharge (an average of 30 days); three-month after onset
  The Perme ICU Mobility Score ranges from 0 to 32 points and is obtained by summing the score of 15 items, each one scored from 2 to 3 points. This score reflects the patient's mobility status in specific circumstances.

SECONDARY OUTCOMES:
The total score-change of the motor domain of the Functional Independence Measure (FIM-motor) | at baseline; at the time of ICU discharge; the time of hospital discharge (an average of 30 days); three-month after onset
  the FIM-motor consist of self-care tasks (eating, grooming, bathing, upper-body dressing, lower-body dressing, and using the toilet), sphincter control (bladder and bowel management), transfers (from bed or a chair to the toilet, bath, or shower), and locomotion ability (walking or wheelchair mobility, and stair climbing)
the achievement level of Modified Trauma ICU Mobility Scale | at baseline; at the time of ICU discharge; the time of hospital discharge
  the achievement of Modified Trauma ICU Mobility Scale, Level 0-10
the days of achievement of the walking motor milestone | up to 3 months
  walking on a level surface for ≥50 meters with or without an assistive device
the values tested by in body s10 about lean body mass parameters | at baseline; at the time of ICU discharge; the time of hospital discharge/ an average of 30 days;
  including phase angle, skeletal muscle mass, body fat mass, total body water etc.
the length of stay in the ICU | up to 3 months
  the length of stay in the ICU
the hospital length of stay | up to 3 months
  the hospital length of stay
the days of ventilator used | up to 3 months
  the days of ventilator used
the discharge disposition after hospital discharge | up to 3 months
  where a patient is being discharged - i.e. home, home with home care, skilled nursing facility, or rehab center.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Chuang, Dr, Principal Investigator — Department of Physical Medicine and Rehabilitation
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yen HC, Chuang HJ, Hsiao WL, Tsai YC, Hsu PM, Chen WS, Han YY. Assessing the impact of early progressive mobilization on moderate-to-severe traumatic brain injury: a randomized controlled trial. Crit Care. 2024 May 22;28(1):172. doi: 10.1186/s13054-024-04940-0. PMID 38778416